CLINICAL TRIAL: NCT05360056
Title: Effect of Continuous Glucose Monitoring Following Hospital Discharge of Patients With Type 2 Diabetes
Brief Title: Continuous Glucose Monitoring Following Hospital Discharge
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathleen Dungan (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Kathleen Dungan, Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021H0426
Record Dates: First submitted 2022-04-26; First posted 2022-05-04 (Actual); Results first posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dexcom CGM (Experimental)
  Interventions: Device: DexCom G6

INTERVENTIONS:
Device: DexCom G6 — Wearable continuous glucose monitor

SUMMARY:
In this 12-week prospective observational cohort study, hospitalized insulin-requiring patients with T2D will receive a Dexcom continuous glucose monitor (CGM) to wear post-hospital discharge. Patients will complete surveys assessing patient-reported outcomes prior to CGM use and following completion of the study. CGM data will be captured by the patient smartphone app and analyzed. Patients will receive personalized CGM targets and alerts for hyperglycemia and hypoglycemia. Customized reports/ decision support will be sent to the usual diabetes provider. The initial observational cohort study design will be followed by an extension phase of 12 weeks in which data on continuation of use and glucose control will be collected but no further reports will be communicated to providers.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Basal insulin use >10 units per day
* Hemoglobin A1c >8.0%
* Smartphone compatible with Clarity App
* Age ≥18 years

Exclusion Criteria:

* Type 1 DM
* Inability to consent
* Pregnancy
* Prisoners
* Discharge to skilled nursing facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Dungan, MD, Principal Investigator — OSU Medical Center
Locations (1):
- The Ohio State University Medical Center - Outpatient Care East, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
• Availability of data and materials: In accordance with institution policy on sharing data and research resources, the final research data from this study may be made available for research purposes under a limited data use agreement specifying criteria for data access, conditions for research use, privacy and confidentiality standards to ensure data security and prohibitions for manipulating data for the purposes of identifying subjects.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexcom CGM
Started | 108
Completed | 66 (primary endpoint, week 12)
Not Completed | 42

BASELINE CHARACTERISTICS:
Arm/Group | Dexcom CGM
Number analyzed (Participants) | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 92
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 106
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 62
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 108
Baseline HbA1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 11.3 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in TIR 70-180 mg/dl
Description: Change in %time in range between 70-180 mg/dl from 2 weeks to 12 weeks.
Time Frame: 12 weeks
Population: 54 participants had data at 2 weeks and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of time spent 70-180 mg/dl
Arm/Group | Dexcom CGM
Number analyzed (Participants) | 54
percentage of time spent 70-180 mg/dl | 8.5 (28)
Statistical Analysis 1: Comparison: Dexcom CGM; Paired t-test was performed comparing the %Time in range from 2 weeks to 12 weeks; Test type: Superiority — paired t-test; p = 0.03, paired t-test — unadjusted p-value; Mean Difference (Net) = 8.51, Standard Deviation 28.0

2. Primary Outcome: % Wear Time >70%
Description: The number of participants with % wear time >70% will be reported.
Time Frame: 12 weeks
Population: 58 participants had CGM wear time at week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Dexcom CGM
Number analyzed (Participants) | 58
Participants | 54

3. Primary Outcome: DTSQc Score
Description: The DTSQc compares the experience of the current treatment with the experience of the treatment before initiation of the study. Scores range from +3 ("much more satisfied now") to -3 ("much less satisfied now"), with 0 (midpoint) representing no change. Higher scores on the DTSQ total score indicate higher treatment satisfaction, and lower scores indicate lower treatment satisfaction. The total score ranges from -18 (maximum deterioration in satisfaction) to +18 (maximum improvement in satisfaction).A score of 0 indicates no change in satisfaction.
Time Frame: 12 weeks
Population: 61 participants had an available DTSQ change score at 12 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dexcom CGM
Number analyzed (Participants) | 61
score on a scale | 8 [6 to 12]
Statistical Analysis 1: Comparison: Dexcom CGM; Test type: Superiority; p < 0.0001, paired Wilcoxon rank test; Wilcoxon signed rank = 9.85

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Sensor adverse events include failure, bleeding, pain, infection and puritus
Arm/Group | Dexcom CGM
All-Cause Mortality (participants affected / at risk) | 1/108
Serious Adverse Events (participants affected / at risk) | 0/108
Other Adverse Events (participants affected / at risk) | 30/108
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexcom CGM (N=108)
Sensor event (Skin and subcutaneous tissue disorders) | 30 (40) — Sensor related events including sensor failure, bleeding, pain, infection, or pruritus

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT05360056/Prot_SAP_001.pdf